CLINICAL TRIAL: NCT04551170
Title: Phase 2 Study of Theophylline Treatment for Pseudohypoparathyroidism
Brief Title: Theophylline Treatment for Pseudohypoparathyroidism - Children 2-12 Years Old
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Ashley Shoemaker, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IND 133103 R01
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Pseudohypoparathyroidism; Albright Hereditary Osteodystrophy; Pseudohypoparathyroidism Type 1a
Keywords: Pseudohypoparathyroidism; PHP; AHO; Albright Hereditary Osteodystrophy
MeSH Terms: conditions — Pseudohypoparathyroidism | interventions — Theophylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Theophylline (Experimental): Theophylline capsules by mouth once daily or Theophylline elixir by mouth q6h (dose determined by serum drug levels)
  Interventions: Drug: Theophylline
- Placebo (Placebo Comparator): Placebo capsule by mouth once daily or Placebo elixir by mouth q6h
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Theophylline — oral theophylline
  Other Names: Theo-24; Elixophyllin
  Arms: Theophylline
Drug: Placebo — Placebo capsule or elixir
  Arms: Placebo

SUMMARY:
Pseudohypoparathyroidism is a genetic disorder with limited treatment options, characterized by early-onset obesity, short stature and resistance to multiple hormones. This phase 2 clinical trial and open-label extension study will test the efficacy of theophylline, a phosphodiesterase inhibitor, in pseudohypoparathyroidism. We hypothesize that theophylline will cause weight loss, slow the rate of growth plate closure and decrease hormone resistance in children.

DETAILED DESCRIPTION:
Pseudohypoparathyroidism (PHP) is a rare, genetic disorder caused by impaired stimulatory G protein (Gsα) signaling through downregulation of the gene, GNAS. The resultant hormone abnormalities can be treated with hormone replacement therapy, but other aspects of the disorder such as early-onset obesity and short stature are without effective treatment options. Gsα signaling is essential for the normal hormonal function of the pituitary, thyroid, gonads, renal proximal tubules and hypothalamus. While many of the resulting hormone deficiencies can be treated with hormone replacement therapy (HRT), HRT is not an effective therapy for the severe early-onset obesity and short stature which are major features of the PHP phenotype. Therefore, the goal of this clinical trial is to test the efficacy of upstream therapy aimed at correcting the function of Gsα-dependent receptors in children with PHP. Gsα-coupled receptor signaling cascade begins with an increase in cyclic adenosine monophosphate (cAMP) which is rapidly degraded by the enzyme phosphodiesterase (PDE). PDE inhibitors act by prolonging cAMP signaling by decreasing the rate of degradation. Given that patients with PHP have reduced, but not completely absent, cAMP production, the investigators seek to test the hypothesis that the PDE inhibitor theophylline will reduce body mass index (BMI), slow the rate of epiphyseal closure, and decrease hormone resistance in children with PHP through improved Gsα-coupled receptor signaling. The investigators will conduct a 52-week randomized, placebo-controlled clinical trial of theophylline in children with PHP. Theophylline is a non-selective PDE inhibitor that is generically available and has a long history of use in pediatric patients, making it an ideal drug for repurposing in youth with PHP. Furthermore, the pharmacokinetics of theophylline are well understood, and serum drug levels are easily measured. Our primary outcome is change in BMI. Secondary outcome measures include change in epiphyseal closure and HRT medication doses.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 to 12 years old
* Clinical diagnosis of PHP (per the EuroPHP network classification guidelines5): Presence of PTH resistance and/or ectopic ossification OR brachydactyly type E plus 2 minor criteria (TSH resistance, other hormonal resistance, developmental delay, intrauterine or post-natal growth retardation, obesity/overweight, specific facial features)
* Obesity (BMI >95th percentile for age/gender and/or ≥30 kg/m2)

Exclusion Criteria:

1. Use of a PDE inhibitor in the past 30 days
2. History of a seizure disorder unrelated to hypocalcemia
3. History of a cardiac arrhythmia (not including bradycardia)
4. Hepatic insufficiency including cirrhosis and acute hepatitis (AST or ALT >3x upper limit of normal)
5. Congestive heart failure
6. Current cigarette use or alcohol abuse
7. Pregnancy or intention to become pregnant during the next year
8. Untreated hypothyroidism (defined as free thyroxine below the lower limit of normal)
9. Active peptic ulcer disease
10. Current use of medications known to effect theophylline levels (see protection of human subjects)
11. History of hypersensitivity to theophylline or other medication components
12. History of Major Depressive Disorder in the past 2 years, lifetime history of suicide attempt, history of any suicidal behavior in the past month, history of other sever psychiatric disorders (e.g. schizophrenia, bipolar disorder)
13. PHQ-9 score is ≥15 or suicidal ideation of type 4 or 5 (C-SSR) in the past month
14. Untreated hypothyroidism or uncontrolled PTH resistance (PTH >2x upper limit of normal), or treatment of these disorders by medications other than calcitriol or levothyroxine (such as Cytomel or Armour thyroid)
15. Unable to comply with study procedures in the opinion of the investigator

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in body mass index | baseline and 52 weeks
  BMI expressed as percent of the 95th percentile

SECONDARY OUTCOMES:
Change in levothyroxine dose | baseline and 52 weeks
  levothyroxine dose (mcg/kg/day)
Change in calcitriol dose | baseline and 52 weeks
  calcitriol dose (mcg/kg/day)
Change in epiphyseal closure | baseline and 52 weeks
  Bone age minus chronologic age

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Shoemaker, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shoemaker AH, Juppner H. Nonclassic features of pseudohypoparathyroidism type 1A. Curr Opin Endocrinol Diabetes Obes. 2017 Feb;24(1):33-38. doi: 10.1097/MED.0000000000000306. PMID 27875418
- [Background] Wang L, Shoemaker AH. Eating behaviors in obese children with pseudohypoparathyroidism type 1a: a cross-sectional study. Int J Pediatr Endocrinol. 2014;2014(1):21. doi: 10.1186/1687-9856-2014-21. Epub 2014 Oct 15. PMID 25337124
- [Background] Mano T, Uchimura K, Hayashi R, Kobahashi T, Fujiwara K, Makino M, Kakizawa H, Nagata M, Nakai A, Wada M, Nagasaka A, Itoh M. Increased urinary phosphate excretion in pseudohypoparathyroidism type II with long-term treatment with phosphodiesterase inhibitor. Horm Metab Res. 1999 Nov;31(11):602-5. doi: 10.1055/s-2007-978804. PMID 10598827
- [Background] Landreth H, Malow BA, Shoemaker AH. Increased Prevalence of Sleep Apnea in Children with Pseudohypoparathyroidism Type 1a. Horm Res Paediatr. 2015;84(1):1-5. doi: 10.1159/000381452. Epub 2015 Apr 23. PMID 25925491
- [Background] Perez KM, Lee EB, Kahanda S, Duis J, Reyes M, Juppner H, Shoemaker AH. Cognitive and behavioral phenotype of children with pseudohypoparathyroidism type 1A. Am J Med Genet A. 2018 Feb;176(2):283-289. doi: 10.1002/ajmg.a.38534. Epub 2017 Nov 28. PMID 29193623
- [Background] Curley KL, Kahanda S, Perez KM, Malow BA, Shoemaker AH. Obstructive Sleep Apnea and Otolaryngologic Manifestations in Children with Pseudohypoparathyroidism. Horm Res Paediatr. 2018;89(3):178-183. doi: 10.1159/000486715. Epub 2018 Feb 16. PMID 29455209
- [Background] Hanna P, Grybek V, Perez de Nanclares G, Tran LC, de Sanctis L, Elli F, Errea J, Francou B, Kamenicky P, Linglart L, Pereda A, Rothenbuhler A, Tessaris D, Thiele S, Usardi A, Shoemaker AH, Kottler ML, Juppner H, Mantovani G, Linglart A. Genetic and Epigenetic Defects at the GNAS Locus Lead to Distinct Patterns of Skeletal Growth but Similar Early-Onset Obesity. J Bone Miner Res. 2018 Aug;33(8):1480-1488. doi: 10.1002/jbmr.3450. Epub 2018 Jun 7. PMID 29693731
- See also: Vanderbilt PHP Research Page — http://www.facebook.com/pseudohypoparathyroidism